CLINICAL TRIAL: NCT02108548
Title: A Phase 1 Ascending Single and Multiple Oral Dose Study to Assess the Safety and Tolerability, Including Gastrointestinal Safety, Pharmacokinetics and Pharmacodynamics of ASP7657 in Caucasian Healthy Male and Female Subjects, Including a Food Effect Cohort
Brief Title: A Study to Assess the Safety and Tolerability, Including Gastrointestinal Safety, Pharmacokinetics and Pharmacodynamics of ASP7657 in Caucasian Healthy Male and Female Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Gastrointestinal safety findings
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 7657-CL-0001; 2013-004357-25 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pharmacokinetics of ASP7657; Pharmacodynamics of ASP7657; Healthy Subjects
Keywords: ASP7657; Pharmacokinetics; Pharmacodynamics; Healthy Subjects; First in man; Safety
MeSH Terms: interventions — ASP7657; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1: ASP7657 Single Ascending Dose (Experimental)
  Interventions: Drug: ASP7657
- Part 1: ASP7657 Single Ascending Dose - Food Effect (Experimental)
  Interventions: Drug: ASP7657
- Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2: ASP7657 Multiple Ascending Dose (Experimental)
  Interventions: Drug: ASP7657
- Part 2: ASP7657 Multiple Ascending Dose Elderly (Experimental)
  Interventions: Drug: ASP7657
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2: Naproxen (Active Comparator)
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: ASP7657 — oral
  Arms: Part 1: ASP7657 Single Ascending Dose; Part 1: ASP7657 Single Ascending Dose - Food Effect; Part 2: ASP7657 Multiple Ascending Dose; Part 2: ASP7657 Multiple Ascending Dose Elderly
Drug: Placebo — oral
  Arms: Part 1: Placebo; Part 2: Placebo
Drug: naproxen — oral
  Arms: Part 2: Naproxen

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple ascending oral doses of ASP7657 in healthy subjects.

DETAILED DESCRIPTION:
Subjects are healthy males aged 18 to 55 years of age (inclusive) (Parts 1 and 2, young cohorts) or the subject is an elderly healthy male or female subject aged 65 years or more (Part 2, elderly cohort).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) range of 18.5 to 30.0 kg/m2, inclusive. The subject weighs at least 50 kg [screening]
* Subject agrees to undergo gastro-duodenoscopy (GDS) if needed (Part 1: in case of gastrointestinal (GI) complaints/positive fecal blood test; Part 2: all subjects)

Exclusion Criteria:

* Subject has known or suspected hypersensitivity to ASP7657 or naproxen, or any components of the formulation used
* Subject has any of the liver function test above the upper limit of normal (ULN)
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Subject has any history or evidence of any clinically significant cardiovascular, GI, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day of admission
* Subject has any clinically significant abnormality
* Subject has a pulse < 40 or > 90 beats per minute (bpm); mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) at day -1. (For elderly subjects the following criteria apply: DBP > 100 mmHg, SBP > 160 mmHg [day of admission])
* Subject has a mean QT interval corrected for heart rate using Fridericia's formula (QTc(F)) of > 430 ms (for males) and > 450 ms (for females).
* Subject uses any prescribed or nonprescribed drugs (including nonsteroidal anti-inflammatory drugs (NSAIDs), anti-coagulants, vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks prior to first study drug administration, except for occasional use of paracetamol (up to 2 g/day)
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of drinking > 21 units (males) or > 14 units (females) of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit or the subject tests positive at screening or clinical admission for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates)
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit
* Subject has significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit regularly
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), anti-hepatitis A virus (HAV) (immunoglobulin [Ig]M), anti-hepatitis C virus (HCV) or anti-human immunodeficiency virus (HIV) 1+2
* Subject has a positive H.Pylori test at screening
* Subject has a positive fecal blood test at screening
* Subject participated in any interventional clinical study or has been treated with any investigational drugs within 90 days or 5 half-lives whichever is longer, prior to the initiation of screening
* Subject is an employee of the Astellas Group or Clinical Research Organization involved in the study
* Subject has a history of peptic ulceration or significant dyspepsia
* Subject uses concomitant medication associated with peptic ulceration, or presence of other risk factors for peptic ulceration
* Subject, if non-elderly, has endoscopic evidence of inflammation, ulceration, erosion, mucosal hemorrhage, or active bleeding in esophagus, stomach, pyloric channel or duodenum, and a mucosal grading scale score > 2 for both stomach and duodenum at baseline visit (Part 2 healthy young male cohorts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Safety assessed by adverse events, vital signs, laboratory tests, electrocardiogram (ECGs), collagen and adenosine diphosphate (ADP)-induced platelet aggregation, and gastrointestinal (GI) safety assessments (Part 2 only) | Up to Day 20

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) profile of ASP7657 after a single dose in plasma: AUCinf, AUClast, tlag, tmax, Cmax, t 1/2, Vz/F, CL/F | Day 1
  Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf), AUC from the time of dosing to the last measurable concentration (AUClast), time prior to the time corresponding to the first measurable (nonzero) concentration (tlag), time of maximum plasma concentration (tmax), maximum plasma concentration (Cmax), terminal elimination half-life (t ½), apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F), and apparent total systemic clearance after single or multiple extravascular dosing (CL/F)
Part 1: PK profile of ASP7657 in urine: Aelast, Aeinf, Aelast%, Aeinf%, CLr | Day 1
  Cumulative amount of drug excreted in urine from time of dosing up to the collection time of the last measurable concentration (Aelast), cumulative amount of drug excreted in urine from time of dosing extrapolated to time infinity (Aeinf), percent of drug dose excreted in urine from time of dosing up to the collection time of the last measurable concentration (Aelast%), percent of drug dose excreted in urine from time of dosing extrapolated to time infinity (Aeinf%), renal clearance (CLr)
Part 1: Pharmacodynamics (PD) profile of tumor necrosis factor alpha (TNF-α) in whole blood: maximum response (Rmax), area under the dose-response curve (AURC), and time to reach maximum response (tmax,R) | Day 1
Part 1: PD in urine: Total urine volume over 24 hours | Day -1 and Day 1
Part 2: PK profile of ASP7657 after first dose in plasma: tlag, tmax, Cmax and AUC from the time of dosing to 24 hours postdose (AUC24) | Day 1
Part 2: PK of ASP7657 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Days 2, 4, 6, 8, 10 and 12
Part 2: PK profile of ASP7657 after last dose in plasma: AUC from the time of dosing to the start of the next dosing interval (AUCtau), tmax, Cmax, t ½, Vz/F, CL/F, Accumulation ration (Racc), peak-trough ratio (PTR) | Day 14
PK profile of ASP7657 after last dose in urine: Aetau, (Aetau%), and CLr | Day 14
  Cumulative amount of drug excreted in urine from the time of dosing to the start of the next dosing interval (Aetau), percent of drug dose excreted in urine over the time interval between consecutive dosing (Aetau%)
Part 2: PD profile of plasma renin activity and aldosterone | Days -1, 7, and 14
Part 2: PD of urine electrolytes: amount excreted over 24 hours (Ae24) | Days -1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, Middlesex, United Kingdom